CLINICAL TRIAL: NCT07169032
Title: The Effect of Er,Cr:YSGG Laser-assisted Topical Anesthetic on Oral Mucosal Anesthesia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Li Zhen Zhong (Other)
Responsible Party: Sponsor-Investigator, Li Zhen Zhong, Master Student, First Affiliated Hospital of Jinan University
Organization: First Affiliated Hospital of Jinan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JNUKY-2023-0149
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Results first posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Anesthesia
Keywords: Er,Cr:YSGG laser; needle-free anesthesia; dental anxiety; oral mucosal anesthesia
MeSH Terms: interventions — Lidocaine; Petrolatum

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Laser + Lidocaine (Experimental): One of three sites in the vestibular groove of the mandibular anterior teeth region of each participant received irradiation with a 2780 nm, 1.0 W Er,Cr:YSGG laser for 1 minute followed by application of 2% lidocaine gel.
  Interventions: Device: Er,Cr:YSGG laser irradiation; Drug: Lidocaine
- Sham Laser + Lidocaine (Sham Comparator): One of three sites in the vestibular groove of the mandibular anterior teeth region of each participant received sham laser irradiation for 1 minute followed by application of 2% lidocaine gel.
  Interventions: Drug: Sham Laser irradiation; Drug: Lidocaine
- Sham Laser + Vaseline (Placebo Comparator): One of three sites in the vestibular groove of the mandibular anterior teeth region of each participant received sham laser irradiation for 1 minute followed by application of Vaseline.
  Interventions: Drug: Sham Laser irradiation; Drug: Vaseline

INTERVENTIONS:
Device: Er,Cr:YSGG laser irradiation — irradiation with a 2780 nm, 1.0 W Er,Cr:YSGG laser for 1 minute
  Arms: Laser + Lidocaine
Drug: Sham Laser irradiation — sham laser irradiation for 1 minute
  Arms: Sham Laser + Lidocaine; Sham Laser + Vaseline
Drug: Lidocaine — 2% lidocaine gel
  Arms: Laser + Lidocaine; Sham Laser + Lidocaine
Drug: Vaseline — Vaseline
  Arms: Sham Laser + Vaseline

SUMMARY:
This study tests whether using an Er,Cr:YSGG laser before applying numbing gel (lidocaine) can help reduce pain during dental procedures compared to traditional methods. Investigators want to know:

Does the laser make the numbing gel work better and longer?

Does it lower pain and keep patients calmer (measured by heart rate)?

Investigators enrolled 20 adults (10 men, 10 women) and assigned them to three groups:

Laser + Numbing Gel: Laser was used on the gums before applying lidocaine.

Sham Laser + Numbing Gel: A fake laser was used with lidocaine.

Sham Laser + Vaseline: A fake laser was used with Vaseline (no numbing effect).

Participants reported pain levels on a scale (0=no pain, 10=worst pain) when a tiny needle touched their gums. Investigators also checked their heart rate.

DETAILED DESCRIPTION:
Participants will be invited to participate in a study observing the anesthetic efficacy of the combination of Er,Cr:YSGG laser and surface anesthetic agent on the oral mucosa. This informed consent form provides participants with detailed information to help participants decide whether to participate in this project. Please read it carefully. If participants have any questions, please raise them to the researcher in charge of the study. Investigators will give participants a comprehensive explanation.

Participants' participation in this study is voluntary. This research has been reviewed by the ethics committee of this research institution.

Research purpose: By measuring the anesthetic depth of the combined use of Er,Cr:YSGG water laser and surface anesthetic agent at different time points in the oral vestibule of the mandibular anterior teeth area, to observe the anesthetic efficacy of the combined use of Er,Cr:YSGG water laser and surface anesthetic agent on the oral mucosa.

Research content and process: Before participants are selected for the study, the doctor will ask about participants basic situation, record participants' medical history, and conduct a routine oral examination. The specific requirements are: no allergy to anesthetic drugs, no mucosal lesions, no pregnancy, no systemic diseases, and good health condition.

If participants' above examinations are qualified, participants will follow the following steps for the study: Rest for half an hour to stabilize blood pressure and heart rate. The nurse will put an electrocardiogram monitor on participants to record the changes in blood pressure and heart rate throughout the process. The doctor will select three sites in the vestibule of the mandibular anterior teeth area and irradiate 1 cm away from the site at a 90-degree angle with water laser or ineffective laser for 1 minute, and then randomly apply lidocaine or vaseline to the three sites. The subjects will not rinse their mouths during the experiment. The doctor will insert an aseptic needle into the mucosa at three sites in the mandibular anterior teeth area 10 minutes, 20 minutes, 30 minutes, 40 minutes and 50 minutes after irradiation, and the subjects will raise their hands to indicate "feeling" or "pain" to stop the needle insertion. The doctor will record the depth of needle insertion.

After the anesthesia, the doctor will check the wound. The doctor will visit the subject's numbness and record the anesthetic duration. Observe whether there are itching, pain, redness and swelling in the wound.

Risks and discomforts: A few people in this clinical experiment may have discomfort symptoms such as itching, pain, and redness. If these discomforts occur, the doctor will handle them promptly. Participants' relevant information will be kept confidential. Investigators will do our best to minimize the possibility of participants' information being exposed.

Benefits of participating in this study: Participants will receive a free panoramic X-ray, full-mouth examination, and supra-gingival scaling.

Cost: The relevant research costs for this project will be borne by the research group. Participants do not need to bear the relevant costs for the research process itself, and it will not increase participants' additional medical treatment costs. If physical harm is caused to participants due to the research itself, the additional medical treatment costs will be compensated or compensated in accordance with relevant national laws and regulations.

As a research subject, participants need to: Provide the true situation of participants' own medical history and current physical condition; Tell the researcher of any discomforts participants experience during this study; Tell the researcher whether participants have participated in other studies recently or are currently participating in other studies, and other matters that may affect the research results or participants' health.

Privacy issue: If participants decide to participate in this study, participants' participation in the trial and participants' personal information during the trial will be kept confidential. Participants' identity information will not be disclosed to members outside the research group unless participants give participants' permission. All research members and the research sponsor are required to keep participants' identity confidential. Participants' file will be stored in a locked filing cabinet and only available for researchers to consult. To ensure the research is conducted in accordance with regulations, when necessary, members of government management departments or ethics review committees will be able to consult participants' personal information at the research institution. When the research results are published, no personal information of participants will be disclosed.

Participants have the right to choose not to participate in this study. During the research process, participants also have the right to withdraw at any time without any reason. Investigators will decide whether the obtained data will be included in the research results according to participants' wishes and the needs of the research. Participants' any rights will not be affected in this case.

If participants need other treatments, or participants fail to follow the research plan, or there is any injury related to the research or any other reasons, the researcher can terminate participants' participation in this study.

Participants can always obtain information about themselves and the progress of this research. If participants have any questions related to this research, or if participants experience any discomfort or injury during the research process, or if participants have any questions regarding the rights of participants in this study, please contact the researcher by phone or other means in a timely manner.

ELIGIBILITY:
Inclusion Criteria:

* could understand and follow given instructions

Exclusion Criteria:

* excessive dental anxiety
* anesthesia allergies
* mucosal lesions
* cardiovascular disease
* diabetes
* pregnancy or lactation
* severe psychiatric disorders
* hearing abnormalities
* speech dysfunction

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Jinan University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Khalighi HR, Mojahedi M, Parandoosh A. Efficacy of Er,Cr:YSGG laser-assisted delivery of topical anesthesia in the oral mucosa. Clin Oral Investig. 2021 Mar;25(3):1055-1058. doi: 10.1007/s00784-020-03399-x. Epub 2020 Jun 18. PMID 32556664

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: site
Period: Overall Study
Arm/Group | Laser + Lidocaine | Sham Laser + Lidocaine | Sham Laser + Vaseline
Started (Note on study design: This study utilized a within-subject, crossover design. All 20 participants received all three interventions (Laser + Lidocaine, Sham Laser + Lidocaine, and Sham Laser + Vaseline) applied to three separate sites in the oral mucosa. Therefore, the number of participants analyzed per group (n=20) is equal to the total number of participants enrolled (N=20). The total number of observations is 60 (20 participants × 3 interventions).) | 20; 20 site | 20; 20 site | 20; 20 site
Completed | 20; 20 site | 20; 20 site | 20; 20 site
Not Completed | 0; 0 site | 0; 0 site | 0; 0 site

BASELINE CHARACTERISTICS:
Units Other Than Participants: site
Groups:
- Total: Total of all reporting groups
Arm/Group | Laser + Lidocaine | Sham Laser + Lidocaine | Sham Laser + Vaseline | Total
Number analyzed (Participants) | 20 | 20 | 20 | 80
Number analyzed (site) | 20 | 20 | 20 | 60
Age, Categorical [Count of Units; unit: site] — Note on study design: This study utilized a within-subject, crossover design. All 20 participants received all three interventions (Laser + Lidocaine, Sham Laser + Lidocaine, and Sham Laser + Vaseline) applied to three separate sites in the oral mucosa. Therefore, the number of participants analyzed per group (n=20) is equal to the total number of participants enrolled (N=20). The total number of observations is 60 (20 participants × 3 interventions).
  site
    number analyzed (Participants) | 20 | 20 | 20 | 20
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 20 | 20 | 20 | 60
    >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Units; unit: site] — Note on study design: This study utilized a within-subject, crossover design. All 20 participants received all three interventions (Laser + Lidocaine, Sham Laser + Lidocaine, and Sham Laser + Vaseline) applied to three separate sites in the oral mucosa. Therefore, the number of participants analyzed per group (n=20) is equal to the total number of participants enrolled (N=20). The total number of observations is 60 (20 participants × 3 interventions).
  site
    number analyzed (Participants) | 20 | 20 | 20 | 20
    Female | 10 | 10 | 10 | 30
    Male | 10 | 10 | 10 | 30
Race (NIH/OMB) [Count of Units; unit: site] — Note on study design: This study utilized a within-subject, crossover design. All 20 participants received all three interventions (Laser + Lidocaine, Sham Laser + Lidocaine, and Sham Laser + Vaseline) applied to three separate sites in the oral mucosa. Therefore, the number of participants analyzed per group (n=20) is equal to the total number of participants enrolled (N=20). The total number of observations is 60 (20 participants × 3 interventions).
  site
    number analyzed (Participants) | 20 | 20 | 20 | 20
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 20 | 20 | 20 | 60
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0
    White | 0 | 0 | 0 | 0
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  number analyzed (Participants) | 20 | 20 | 20 | 20
  China | 20 | 20 | 20 | 20

OUTCOME MEASURES:

1. Primary Outcome: Insertion Depth at Initial Sensory Detection
Description: Insert a sterile needle into the mucosa at the sites. Record the Insertion depth when participants perceived an "initial sensory detection"
Time Frame: 10, 20, 30, 40, and 50 minutes
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Laser + Lidocaine | Sham Laser + Lidocaine | Sham Laser + Vaseline
Number analyzed (Participants) | 20 | 20 | 20
mm
  10 min | 7.75 (4.35) | 4.65 (3.10) | 0.4 (1.34)
  20 min | 8.55 (5.40) | 5.45 (3.72) | 0.41 (1.35)
  30 min | 9.28 (7.07) | 3.99 (4.40) | 0.38 (1.34)
  40 min | 4.40 (4.89) | 1.79 (2.74) | 0.375 (1.34)
  50 min | 2.56 (3.60) | 1.44 (3.50) | 0.52 (2.01)

2. Primary Outcome: Insertion Depth at Pain
Description: Insert a sterile needle into the mucosa at the sites. Record the Insertion depth when participants felt "pain".
Time Frame: 10, 20, 30, 40, and 50 minutes
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Laser + Lidocaine | Sham Laser + Lidocaine | Sham Laser + Vaseline
Number analyzed (Participants) | 20 | 20 | 20
mm
  10 min | 12.30 (5.42) | 8.20 (3.58) | 1.17 (2.60)
  20 min | 14.70 (6.51) | 9.15 (3.90) | 1.15 (2.72)
  30 min | 15.45 (6.79) | 7.46 (5.22) | 0.76 (1.78)
  40 min | 10.25 (5.93) | 4.84 (4.19) | 1.13 (2.40)
  50 min | 5.46 (4.87) | 2.72 (4.76) | 0.95 (2.47)

3. Primary Outcome: Pain Score at Initial Sensory Detection
Description: Insert a sterile needle into the mucosa at the sites. Record the pain score when participants perceived an "initial sensory detection". Evaluated with a linear visual analog scale. "0" represents no pain, and "10" represents the most intense pain imaginable.
Time Frame: 10, 20, 30, 40, and 50 minutes
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Laser + Lidocaine | Sham Laser + Lidocaine | Sham Laser + Vaseline
Number analyzed (Participants) | 20 | 20 | 20
Units on a Scale
  10 min | 0.65 (0.34) | 0.90 (0.39) | 1.27 (0.77)
  20 min | 0.75 (0.62) | 1.07 (0.60) | 1.07 (0.74)
  30 min | 0.64 (0.35) | 0.95 (0.56) | 1.18 (0.83)
  40 min | 0.61 (0.35) | 0.92 (0.55) | 1.03 (0.80)
  50 min | 0.75 (0.43) | 0.93 (0.59) | 1.07 (0.74)

4. Primary Outcome: Pain Score at Pain
Description: Insert a sterile needle into the mucosa at the sites. Record the pain score when participants felt "pain". Evaluated with a linear visual analog scale. "0" represents no pain, and "10" represents the most intense pain imaginable.
Time Frame: 10, 20, 30, 40, and 50 minutes
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Laser + Lidocaine | Sham Laser + Lidocaine | Sham Laser + Vaseline
Number analyzed (Participants) | 20 | 20 | 20
Units on a Scale
  10 min | 1.45 (0.75) | 1.79 (0.84) | 2.77 (2.99)
  20 min | 1.37 (0.71) | 1.69 (0.76) | 1.81 (0.82)
  30 min | 1.22 (0.66) | 1.64 (0.84) | 1.87 (0.97)
  40 min | 1.21 (0.64) | 1.67 (0.78) | 1.80 (0.91)
  50 min | 1.35 (0.68) | 1.58 (0.73) | 1.79 (0.81)

5. Primary Outcome: Heart Rate
Description: Insert a sterile needle into the mucosa at the sites. Record the heart rate with an electrocardiogram monitor when participants felt "pain".
Time Frame: 10, 20, 30, 40, and 50 minutes
Measure: Mean (Standard Deviation); unit: BPM
Arm/Group | Laser + Lidocaine | Sham Laser + Lidocaine | Sham Laser + Vaseline
Number analyzed (Participants) | 20 | 20 | 20
BPM
  10 min | 66.75 (7.48) | 75.35 (7.22) | 75.85 (9.02)
  20 min | 65.95 (7.92) | 74.20 (9.16) | 76.15 (10.30)
  30 min | 65.05 (7.54) | 74.45 (9.17) | 75.60 (8.89)
  40 min | 66.40 (7.74) | 74.20 (9.89) | 76.95 (8.40)
  50 min | 65.70 (7.40) | 74.10 (8.90) | 76.80 (9.33)

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, up to 1 week
Arm/Group | Laser + Lidocaine | Sham Laser + Lidocaine | Sham Laser + Vaseline
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT07169032/Prot_SAP_001.pdf
  • Informed Consent Form (2023-12-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT07169032/ICF_002.pdf